CLINICAL TRIAL: NCT00324597
Title: A Phase Ib, Open-Label, Sequential, Dose-Finding, Study of AMG 706 in Combination With Gemcitabine to Treat Subjects With Solid Tumors
Brief Title: AMG 706 and Gemcitabine in Treating Patients With Advanced Solid Tumors or Lymphoma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000481095; UCLA-0506055-01
Record Dates: First submitted 2006-05-10; First posted 2006-05-11 (Estimated); Last update posted 2013-09-17 (Estimated); Status verified 2007-04

CONDITIONS: Lung Cancer; Lymphoma; Lymphoproliferative Disorder; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific; recurrent adult grade III lymphomatoid granulomatosis; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage III mantle cell lymphoma; stage IV mantle cell lymphoma; stage III marginal zone lymphoma; stage IV marginal zone lymphoma; stage III small lymphocytic lymphoma; stage III cutaneous T-cell non-Hodgkin lymphoma; stage IV cutaneous T-cell non-Hodgkin lymphoma; stage III adult T-cell leukemia/lymphoma; recurrent adult Hodgkin lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent adult T-cell leukemia/lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent mantle cell lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; splenic marginal zone lymphoma; stage III adult Burkitt lymphoma; stage III adult diffuse large cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage III adult Hodgkin lymphoma; stage III adult immunoblastic large cell lymphoma; stage III adult lymphoblastic lymphoma; Waldenström macroglobulinemia; recurrent mycosis fungoides/Sezary syndrome; stage III mycosis fungoides/Sezary syndrome; stage IV mycosis fungoides/Sezary syndrome; stage IV adult Burkitt lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult Hodgkin lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV adult T-cell leukemia/lymphoma; adenocarcinoma of the lung; bronchoalveolar cell lung cancer; large cell lung cancer; stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer; recurrent adult Burkitt lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse small cleaved cell lymphoma; stage IV small lymphocytic lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; anaplastic large cell lymphoma; angioimmunoblastic T-cell lymphoma; post-transplant lymphoproliferative disorder; recurrent non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Lymphoma; Lymphoproliferative Disorders; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, T-Cell, Cutaneous; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Hodgkin Disease; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Waldenstrom Macroglobulinemia; Mycosis Fungoides; Sezary Syndrome; Adenocarcinoma of Lung; Adenocarcinoma, Bronchiolo-Alveolar; Carcinoma, Non-Small-Cell Lung; Lymphoma, Large-Cell, Anaplastic; Immunoblastic Lymphadenopathy | interventions — Gemcitabine; motesanib diphosphate

INTERVENTIONS:
Drug: gemcitabine hydrochloride
Drug: motesanib diphosphate
Other: pharmacological study

SUMMARY:
RATIONALE: AMG 706 may stop the growth of cancer cells by blocking blood flow to the cancer or by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as gemcitabine, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving AMG 706 together with gemcitabine may kill more cancer cells.

PURPOSE: This phase I trial is studying the side effects and best dose of AMG 706 when given together with gemcitabine in treating patients with advanced solid tumors or lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the maximum tolerated dose and safety of AMG 706 when given in combination with gemcitabine hydrochloride in patients with advanced solid tumors or lymphoma.

Secondary

* Determine the pharmacokinetic profiles of this regimen in these patients.

OUTLINE: This is a multicenter, open-label, dose-escalation study of AMG 706.

Patients receive oral AMG 706 once daily on days 2-56 and gemcitabine hydrochloride IV over 30 minutes on days 1, 8, 15, 22, 29, 36, and 43 of course 1. For all subsequent courses, patients receive oral AMG 706 on days 1-28 and gemcitabine hydrochloride IV over 30 minutes on days 1, 8, and 15. Treatment repeats every 4 weeks for up to 10 courses in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of AMG 706 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 3 of 6 patients experience dose-limiting toxicity.

During the first course of study treatment, patients undergo blood collection periodically for pharmacokinetic analysis.

After completion of study treatment, patients are followed periodically for up to 5 years.

PROJECTED ACCRUAL: Approximately 18 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed advanced solid tumors or lymphoma
* Must have measurable disease outside a previously irradiated field OR regrowth of tumor within a previously irradiated field
* Must be a candidate for gemcitabine hydrochloride treatment, in the opinion of the investigator
* No untreated or symptomatic brain metastases
* No tumors with direct bowel invasion
* No other hematological malignancies
* No non-small cell lung cancer of squamous cell histology or large central tumor (lesions ≥ 3 cm and located adjacent to or within the hilum or mediastinum)

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Not pregnant
* No nursing during and for 6 months after completion of study treatment
* Fertile patients must use effective contraception during and for 6 months after completion of study treatment
* Negative pregnancy test
* Able to swallow oral medication
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 9 g/dL
* Creatinine ≤ 2.0 mg/dL OR creatinine clearance ≥ 40 mL/min
* Albumin-adjusted calcium ≥ 8 mg/dL
* Urine protein < 30 mg/dL by urinalysis or < 1+ by dipstick OR < 500 mg by 24-hour urine collection
* AST or ALT ≤ 2.5 times upper limit of normal (ULN) (5.0 times ULN in the presence of liver metastasis or primary hepatic neoplasm)
* Bilirubin ≤ 2 times ULN
* PT ≤ 2.0
* INR or PTT ≤ 1.5 times ULN
* Systolic blood pressure (BP) ≤ 145 mm Hg and diastolic BP ≤ 85 mm Hg (stable antihypertensive medication allowed)
* No myocardial infraction within the past year
* No arterial thrombosis or deep vein thrombosis within the past year
* No unstable angina
* No congestive heart failure
* No New York Heart Association class III-IV cardiac disease
* No other unstable or uncontrolled disease or condition relating to or impacting cardiac function
* No HIV positivity
* No other condition that would preclude study participation, compliance, or follow-up assessments

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior enrollment into this study
* At least 1 month since prior investigational device or drug trial
* At least 1 month since prior major surgical procedure
* At least 3 weeks since prior systemic chemotherapy
* At least 2 weeks since prior radiotherapy
* At least 2 weeks since prior rifampin or phenobarbital
* At least 1 week since prior treatment with any of the following:

  * Ketoconazole
  * Itraconazole
  * Clarithromycin
  * Erythromycin
  * Cyclosporine or tacrolimus
  * Nefazodone
  * Herbal medications containing Hypericum perforatum (St. John's wort)
* At least 1 week since prior and no concurrent warfarin

  * Concurrent prophylactic anticoagulation therapy (e.g., low-dose warfarin [≤ 2 mg/day] or low molecular weight heparin) for venous or arterial access devices allowed
* No prior or concurrent kinase insert domain-receptor inhibitors
* No concurrent chemotherapy, radiotherapy, hormone-directed cancer therapy, or tumor-directed antibody therapy

  * Gonadotropin releasing-hormone agonist therapy allowed
* No concurrent interferon
* No concurrent grapefruit juice or whole grapefruit
* No other concurrent standard or investigational drugs or antitumor treatment, including c-kit, platelet-derived growth factor, vascular endothelial growth factor, or epidermal growth factor inhibitors
* No elective surgery during or for 2 weeks after completion of the last dose of AMG 706

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2005-10

PRIMARY OUTCOMES:
Incidence of dose-limiting toxicity as assessed by NCI CTCAE v3.0
Maximum tolerated dose as assessed by NCI CTCAE v3.0

SECONDARY OUTCOMES:
Pharmacokinetic profiles as measured by blood sampling at weeks 1, 2, 9, 13, 21, 29, 37, 45, and 49
Incidence of adverse events, serious adverse events, and laboratory abnormalities not defined as dose-limiting toxicities as assessed by NCI CTCAE v3.0
Response rate (complete and partial response) as measured by modified RECIST at weeks 12, 24, 36, 48, and 49
Biomarkers as measured by RNA transcript profiling and/or proteomic methods at weeks 1, 2, 4, 9, 13, 21, 29, 37, 45, 49

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn Britten, MD, Principal Investigator — Jonsson Comprehensive Cancer Center
Locations (1):
- Jonsson Comprehensive Cancer Center at UCLA, Los Angeles, California, United States